CLINICAL TRIAL: NCT00828282
Title: High-dose HMG-CoA Inhibitor Simvastatin for Patients With Relapsed CLL: Pilot Trial and Pharmacokinetic-pharmacodynamic Studies
Brief Title: High-dose HMG-CoA Inhibitor Simvastatin Relapsed CLL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: John Haslip (Other)
Responsible Party: Sponsor-Investigator, John Haslip, Director, Clinical Research and Data Management Shared Resource Facility, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-LEUK-06-MCC
Record Dates: First submitted 2009-01-22; First posted 2009-01-23 (Estimated); Last update posted 2014-05-26 (Estimated); Status verified 2014-05

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Chronic Lymphocytic Leukemia; Simvastatin; Zocor
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Simvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Simvastatin

INTERVENTIONS:
Drug: Simvastatin — Treatment will be administered on an outpatient basis. Subjects will be given 7.5 mg/kg twice daily of Simvastatin for 7 days on a 21-day cycle with a goal of 6 cycles.
  Other Names: Zocor

SUMMARY:
The primary aim of this trial is to generate a preliminary analysis of this novel therapeutic approach and laboratory studies for patients with recurrent or refractory CLL. Further, this pilot trial will demonstrate the feasibility of the translational science methods proposed for this new collaboration of investigators. The investigators hypothesize that patients with relapsed CLL are recruitable to this study, that the methods for measuring simvastatin concentration and target protein translation are feasible, and that the investigators can efficiently apply the laboratory research methods to patient blood samples before and after patients have taken the study medication.

ELIGIBILITY:
Eligibility Criteria:

* Patients must have histologically or cytologically confirmed chronic lymphocytic leukemia (CLL). Criteria for diagnosis are as per the WHO classification of hematologic tumors (Jaffe 2001). As per the 1996 NCI guidelines for CLL "[second-line or later] treatment of CLL is generally palliative in intent; therefore, patients who have relapsed may be followed without therapy until they experience disease-related symptoms or progressive disease, with deterioration of blood counts, discomfort from lymphadenopathy or hepatosplenomegaly, recurrent infections, or associated autoimmune disorders" (Cheson 1996).
* Age >18 years. Because no dosing or adverse event data are currently available on the use of high-dose simvastatin in patients <18 years of age, children are excluded from this study.
* Life expectancy of greater than 6 months.
* ECOG performance status #2 or better.
* Patients must have normal organ and marrow function as defined below:

  * total bilirubin within normal institutional limits unless resulting from documented hemolysis
  * AST(SGOT)/ALT(SGPT) ≤1.5 X institutional upper limit of normal
  * creatinine ≤ 1.5 institutional upper limit of normal OR
  * creatinine clearance >60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal
  * Creatine phosphokinase ≤ 1.5 institutional upper limit of normal
* Patients with active infections requiring systemic antibiotics should be excluded until resolution of infection
* The effects simvastatin on the developing human fetus at the studied therapeutic dose are unknown. For this reason and because HMG-CoA reductase inhibitors may be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
* Patients may not be receiving any other investigational agents.
* Patients with known brain or nervous system disease should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to simvastatin.
* Patients receiving any medications or substances that are inhibitors or inducers of CYP3A4 are ineligible. Lists including medications and substances known or with the potential to interact with the CYP3A4 isoenzymes are provided in the appendix.
* Patients may not take other anti-cholesterol treatments during this study. Patients who were previously taking anti-cholesterol treatment prior to study entry must be off the anti-cholesterol medications for 14 days before enrolling on this trial.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, diarrhea, myopathy, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because HMG-CoA reductase inhibitors are a drug class with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with simvastatin, breastfeeding should be discontinued if the mother is treated with simvastatin.
* HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with simvastatin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2009-03; Primary Completion 2011-01 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Evaluate the feasibility of investigators to recruit, retain & evaluate responses in a pilot study of participants with relapsed/refractory CLL treated with 7.5 mg/kg of simvastatin taken orally twice daily on days 1-7 of every 21 day cycles for 6 cycles | Begining of therapy and followed for 2 years after completing therapy
Evaluate the feasibility of the proposed methods to determine the plasma and intra-cellular pharmacokinetics after high-dose simvastatin | During therapy
Evaluate the feasibility of proposed methods to determine if high-dose simvastatin treatment affects the prenylation dependent cellular localization of Rho GTPase proteins and to assess the apoptotic index of CLL cells from treated participants | During therapy
Evaluate the feasibility of proposed methods to identify changes in gene expression following high-dose simvastatin treatment | Druing treatment

CONTACTS AND LOCATIONS:
Overall Officials: John Hayslip, MD, MSCR, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

REFERENCES:
- See also: Markey Cancer Center Blood and Marrow Transplant Study Search — http://markey.uky.edu/studysearch/default.aspx?site=Blood%20and%20Marrow%20Transplant